CLINICAL TRIAL: NCT05934695
Title: The Impact of Lymphedema Severity on Shoulder Joint Function and Muscle Activation Patterns in Breast Cancer Survivors: A Cross-Sectional Study
Brief Title: Lymphedema Severity on Shoulder Joint Function and Muscle Activation Patterns in Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 010/28202306
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Breast Cancer Female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild lymphedema (stage 1): International Society of Lymphology lymphedema severity stage 1, characterized by swelling with pitting, normal skin and tissue turgor. Participants assigned to this group will have mild swelling and tightness of the arm.
  Interventions: Other: Lymphedema severity stratification
- Moderate lymphedema (stage 2): International Society of Lymphology lymphedema severity stage 2, characterized by swelling with pitting as well as skin and tissue changes such as dermal thickening. Participants assigned to this group will have moderate swelling and tightness of the arm as well as skin changes without distortional warty-overgrowth or elephantiasis folds.
  Interventions: Other: Lymphedema severity stratification
- Severe lymphedema (stage 3): International Society of Lymphology lymphedema severity stage 3, characterized by swelling with non-pitting, and warty-overgrowth or elephantiasis folds of skin. Participants assigned to this group will have severe swelling and tightness of the arm with warty overgrowth of skin.
  Interventions: Other: Lymphedema severity stratification

INTERVENTIONS:
Other: Lymphedema severity stratification — Participants will be stratified into one of three lymphedema severity groups based on the International Society of Lymphology lymphedema severity staging:
  Mild (stage 1): swelling with pitting; normal skin and tissue turgor Moderate (stage 2): swelling with pitting; dermal thickening; skin changes without distortional warty-overgrowth Severe (stage 3): swelling with non-pitting; warty overgrowth or elephantiasis folds

SUMMARY:
Breast cancer-related lymphedema (BCRL) is a common complication affecting the upper extremity following breast cancer treatment. This study aims to investigate the relationship between lymphedema severity and shoulder joint function and muscle activation patterns in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Adults (18 years or older)
* Diagnosis of breast cancer-related lymphedema for a minimum of 3 months
* No current evidence of active cancer
* Able to provide informed consent

Exclusion Criteria:

* Pre-existing musculoskeletal conditions affecting the upper extremities (e.g. adhesive capsulitis, rotator cuff tear)
* Previous upper extremity surgery
* Physical inability to perform the required physical movements and assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to recruit women with different severity levels of breast cancer-related lymphedema, an upper limb condition that can result from breast cancer treatment causing swelling and other impairments. By assessing women at different points along the continuum of lymphedema severity, the impact of severity on shoulder function and related outcomes can be examined.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Shoulder joint mobility | baseline
  shoulder flexion, abduction, external rotation and extension range of motion measured using a digital inclinometer.
Muscle activation patterns (Amplitude) | baseline
  Surface EMG recording of muscle activation patterns (amplitude) of the biceps brachii, anterior/middle/posterior deltoid, pectoralis major and latissimus dorsi during shoulder elevation. Amplitude will be reported in units of microvolts (µV)
Muscle activation patterns (Timing) | baseline
  Surface EMG recording of muscle activation patterns (timing) of the biceps brachii, anterior/middle/posterior deltoid, pectoralis major and latissimus dorsi during shoulder elevation. Timing will be reported in units of milliseconds (ms).

SECONDARY OUTCOMES:
Shoulder flexors strength | baseline
  Maximal shoulder flexor abductor strength measured as force production (N) using a handheld dynamometer. The average of 3 trials for each muscle group will be calculated.
Shoulder abductor strength | baseline
  Maximal shoulder abductor strength measured as force production (N) using a handheld dynamometer. The average of 3 trials for each muscle group will be calculated.
Self-reported upper extremity function | baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, developed by the Institute for Work and Health, is used to measure patient-reported functional outcomes. The DASH questionnaire consists of 30 questions regarding limitations to complete physical activities due to upper extremity pain/impairment. Participants will be asked to respond to each question based on their experiences over the preceding week according to a 5-point Likert scale ranging from 1 (no difficulty) to 5 (unable to do). Responses will be scored out of 5 and averaged to produce a score out of 100 with higher scores representing greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No